CLINICAL TRIAL: NCT06914232
Title: Efficacy of Warm Compress Therapy in Enhancing Tear Film Quality and Reducing Postoperative Dry Eye Syndrome After Cataract Surgery: A Randomized Controlled Trial
Brief Title: Efficacy of Warm Compress Therapy in Enhancing Tear Film Quality and Reducing Postoperative DES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/817
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Compress (Experimental)
  Interventions: Combination Product: Warm Compress
- Standard Care (Active Comparator)
  Interventions: Diagnostic Test: Standard Care

INTERVENTIONS:
Combination Product: Warm Compress — The intervention involves perioperative Warm compress therapy administered to the participants in the intervention group before and after cataract surgery for 3 seesions per week for 6 weeks. The therapy aims to enhance tear film stability and alleviate symptoms of dry eye by delivering warm compress to the meibomian glands to restore their function. Participants will undergo a session of warm compress therapy prior to surgery and another one following the surgery.
  Arms: Warm Compress
Diagnostic Test: Standard Care — The control group will receive standard care, which includes artificial tears or other conventional methods for dry eye management for 3 sessions per week for 6 weeks. , but they will not receive Warm Compress therapy.
  Arms: Standard Care

SUMMARY:
Dry eye disease (DED) is a multifactorial condition often exacerbated by cataract surgery, leading to discomfort and visual disturbances. Meibomian gland dysfunction (MGD), a key cause of DED, contributes to tear film instability, which can be managed with warm compress therapy.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of perioperative warm compress therapy (TPT) in improving tear film stability and reducing dry eye symptoms following cataract surgery. This randomized controlled trial (RCT) will involve 54 patients with estimated attrition rate 60 participants aged 50-70 with moderate to severe dry eye symptoms and tear film instability, as indicated by high Ocular Surface Disease Index (OSDI) scores. Participants will be randomly assigned to either an intervention group, receiving warm compress therapy before and after surgery, or a control group receiving standard dry eye treatments for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 to 70 years
* Patients scheduled for cataract surgery (both unilateral and bilateral).
* Patients with preoperative moderate to severe dry eye symptoms, which will be assessed using the Ocular Surface Disease Index (OSDI).

Exclusion Criteria:

* Patients with OSDI, indicating severe dry eye disease which suggests severe dry eye disease. These patients might require more intensive treatments beyond Warm Compress therapy.
* Patients with systemic diseases (e.g., rheumatoid arthritis, lupus) that affect tear production or who are using medications that severely reduce tear production (e.g., chronic use of antihistamines or systemic corticosteroids).
* Patients with significant pre-existing corneal pathology (e.g., corneal dystrophies, corneal scars) that could affect the results of cataract surgery or thermal pulsation therapy.
* Patients with active ocular infections (e.g., conjunctivitis, keratitis) or inflammation at the time of screening or surgery.
* Patients with a history of previous ocular surgeries (excluding cataract surgery) in the study eye, such as refractive surgery (LASIK, PRK) or corneal transplants.
* Patients with a known allergy or contraindication to Warm Compress therapy or its components.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 12 Months
  The Ocular Surface Disease Index (OSDI) is a 12-question questionnaire used to assess the severity of dry eye symptoms and their impact on vision-related function, scored on a scale of 0 to 100, with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hakeem mahmood trust hospital address alam chowk mean baipas, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No